CLINICAL TRIAL: NCT04816955
Title: Dietary Recommendations for Reducing Free Sugar Intakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PhDBoxall
Record Dates: First submitted 2021-03-17; First posted 2021-03-25 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Dietary Recommendations
Keywords: free sugars; dietary intake; dietary recommendations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator, all researchers and analysts will be blinded to treatment. Participants can not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutrient-based recommendations (Experimental): Participants in this group will be given nutrient-based recommendations to reduce free sugar intakes.
  Interventions: Behavioral: Dietary recommendations
- Nutrient- and food-based recommendations (Experimental): Participants in this group will be given nutrient- and food-based recommendations to reduce free sugar intakes.
  Interventions: Behavioral: Dietary recommendations
- Nutrient- and food-based recommendations with food swaps (Experimental): Participants in this group will be given nutrient- and food-based recommendations and advice on food swaps to reduce free sugar intakes.
  Interventions: Behavioral: Dietary recommendations
- Control (Placebo Comparator): Participants in this group will not be given any recommendations to reduce free sugar intakes.
  Interventions: Behavioral: Dietary recommendations

INTERVENTIONS:
Behavioral: Dietary recommendations — Dietary recommendations, with increasing additional behavioural/practical advice or no dietary recommendations

SUMMARY:
This randomised controlled trial aims to assess the impacts of the current recommendations by Public Health England for reducing free sugar intakes, on total energy intakes of free sugar in a sample of the UK population.

DETAILED DESCRIPTION:
The primary objective of this randomised control trial is to assess the impacts of Public Health England's (PHE) current free sugar reducing advice, for reducing total energy intakes (TEI) of free sugar. A total of 240 participants (age 18-65years) consuming diets >5% total energy intake from dietary free sugars will be recruited from across the Dorset region. Participants to be randomly assigned into the following recommendation interventions groups: 1) Reduce free sugar intake to <5% TEI (nutrient-based recommendations); 2) Reduce free sugar intake to <5% TEI, via reducing intake of specific foods identified as high in free sugars (nutrient- + food-based recommendations); 3) Reduce free sugar intake to <5% TEI, via reducing intake of specific foods identified as high in free sugars and replace/swap with low sugar versions (nutrient- + food-based recommendations with swaps); and 4) Control Group. The primary outcome will be changes in free sugar consumption from baseline to endpoint at week 12. Secondary outcomes include change in: BMI; dietary profiles; sweetness preference; sweetness liking; food choices; low calorie sweetener intakes and adherence levels.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years;
* able to provide consent and complete all study materials;
* consuming >5% of TEI from free sugars; and
* residing in the South of England.

Exclusion criteria:

* individuals who are pregnant or breastfeeding;
* underweight (BMI <18.5);
* have pre-existing medical conditions affecting swallow ability, taste and smell perception;
* currently or within 3 months of starting the study are following a specific dietary programme (e.g.: Slimming World);
* current smokers or have smoked within 3 months of the study start date;
* have pre-existing clinical conditions such as diabetes mellitus, eating disorders, Crohn's disease and other illness's leading to participants receiving external nutritional advice and dietary restrictions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Appleton, Principal Investigator — Bournemouth University
Locations (1):
- Bournemouth University, Bournemouth, US and Canada Only, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data will be available on completion of the trial from the PI
Supporting Information: Study Protocol, SAP
Time Frame: On study completion

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
Started | 61 | 60 | 63 | 58
Completed | 52 | 53 | 54 | 41
Not Completed | 9 | 7 | 9 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control | Total
Number analyzed (Participants) | 61 | 60 | 63 | 58 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (14) | 38.3 (12.2) | 42.5 (13.4) | 41.7 (12.6) | 41.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 55 | 53 | 214
  Male | 7 | 8 | 8 | 5 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 53 | 50 | 58 | 51 | 212
  Other background | 8 | 10 | 5 | 7 | 30
Region of Enrollment [Number; unit: participants]
  United Kingdom | 61 | 60 | 63 | 58 | 242
Free sugar intakes [Mean (Standard Deviation); unit: percentage of total energy intake] | 10.1 (5.2) | 10.7 (4.8) | 10.2 (4.4) | 10.4 (5.1) | 10.3 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Free Sugar Intakes
Description: Percentage energy intake from free sugars, assessed using diet diaries
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Error); unit: percentage of total energy intake
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
Number analyzed (Participants) | 61 | 60 | 63 | 58
percentage of total energy intake | 7.7 (0.7) | 7.4 (0.7) | 7.1 (0.6) | 9.2 (0.7)

2. Primary Outcome: Number of Participants Who Adhered to the Recommendations Provided
Description: Adherence to the recommendations provided, assessed using diet diaries and self-reported adherence
Time Frame: 12 weeks from baseline
Measure: Number; unit: participants
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
Number analyzed (Participants) | 61 | 60 | 63 | 58
participants | 38 | 39 | 39 | 25

3. Secondary Outcome: Dietary Intakes
Description: Energy intake, assessed using diet diaries
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
Number analyzed (Participants) | 61 | 60 | 63 | 58
kcal/day | 1512 (60) | 1466 (70) | 1495 (56) | 1516 (56)

4. Secondary Outcome: BMI
Description: Body Mass Index, assessed using researcher measurements or researcher-observed self-measurements
Time Frame: 12 weeks from baseline
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
Number analyzed (Participants) | 61 | 60 | 63 | 58
kg/m2 | 27.2 (0.7) | 28.1 (0.7) | 27.1 (0.7) | 27.4 (0.8)

5. Secondary Outcome: Sweet Food Preferences
Description: Preferences for various sweet foods/fluids, assessed using a taste test, where participants sample several sweet and non-sweet foods and rate them for pleasantness on a 100mm Visual Analogue Scale. Higher scores signify stronger preferences
Time Frame: 12 weeks from baseline
Reporting Status: Not Posted

6. Secondary Outcome: Sweet Food Choices
Description: Selection of sweet foods/fluids at a given meal, assessed where participants can consume freely from a meal composed of sweet and non-sweet foods, and proportion of sweet foods consumed is measured in terms of weight consumed
Time Frame: 12 weeks from baseline
Reporting Status: Not Posted

7. Secondary Outcome: Sweet Food Attitudes
Description: Attitudes towards sugar, sweeteners, and sweet-tasting foods, assessed using a questionnaire, soon to be published. Higher scores denote stronger attitudes.
Time Frame: 12 weeks from baseline
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Adverse events, assessed by self-report
Time Frame: Baseline to 12 weeks
Measure: Number; unit: participants
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
Number analyzed (Participants) | 61 | 60 | 63 | 58
participants | 1 | 1 | 2 | 1

9. Secondary Outcome: Eating-based Attitudes
Description: Attitudes towards eating, assessed using the Three Factor Eating Questionnaire (Karlsson J, et al. IJO 2000; 24: 1715-1725)
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Eating-based Motivations
Description: Motivations towards eating, assessed using the Food Choice Questionnaire (Steptoe et al., Appetite 1995, 25(3): 267-84). Higher scores denote stronger motivations
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Quality of Life (Subjective Wellbeing)
Description: Quality of Life, measured using the SF-36 questionnaire (Ware et al, 1996), where Quality of Life is assessed out of 100, where a higher score demonstrates better quality of life
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Self-report
Arm/Group | Nutrient-based Recommendations | Nutrient- and Food-based Recommendations | Nutrient- and Food-based Recommendations With Food Swaps | Control
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60 | 0/63 | 0/58
Serious Adverse Events (participants affected / at risk) | 1/61 | 1/60 | 2/63 | 1/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60 | 0/63 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nutrient-based Recommendations (N=61) | Nutrient- and Food-based Recommendations (N=60) | Nutrient- and Food-based Recommendations With Food Swaps (N=63) | Control (N=58)
Adverse event (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) — Details not requested

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT04816955/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT04816955/SAP_000.pdf